CLINICAL TRIAL: NCT00037375
Title: Physical Activity, Body Composition, and Prevalent Asthma
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1166; R03HL068245 (NIH)
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-02

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To investigate the relationship of childhood lifestyle and physical characteristics to prevalent asthma.

DETAILED DESCRIPTION:
BACKGROUND:

Morbidity and mortality from pediatric asthma have been increasing in developed countries over the past three decades, making asthma the most common chronic disease of children. A joint session at the American Thoracic Society meeting in May 2000 was titled "Childhood Asthma: Is Change in Lifestyle the Key"? During this session, the hypothesis was advanced that a lack of physical exercise and higher levels of childhood obesity may be contributing to an increased incidence of asthma among United States children.

DESIGN NARRATIVE:

Data from physician diagnosed pediatric asthma were assessed for relationships with the potential risk factors body mass index, percent fat and lean tissue, obesity, and physical activity. The data pertained to a large population-based multi-ethnic cohort of school children (n=826) from the Detroit area for whom, using dual-energy x-ray absorptiometry, precise measurements of whole body bone mass, and soft tissue composition were collected along with height and weight measurements in 1992-1993, when the children were nine years old. Detailed data on physical activity, collected with consultation with an exercise physiologist, and prevalent asthma diagnosis and symptoms, collected under the direction of a respiratory disease/pediatric epidemiologist and a pediatric allergist, were obtained at the same time.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-07; Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Peterson — Case Western Reserve University

REFERENCES:
- [Background] Johnson CC, Ownby DR, Zoratti EM, Alford SH, Williams LK, Joseph CL. Environmental epidemiology of pediatric asthma and allergy. Epidemiol Rev. 2002;24(2):154-75. doi: 10.1093/epirev/mxf013. No abstract available. PMID 12762090
- [Background] Alford SH, Zoratti E, Peterson EL, Maliarik M, Ownby DR, Johnson CC. Parental history of atopic disease: disease pattern and risk of pediatric atopy in offspring. J Allergy Clin Immunol. 2004 Nov;114(5):1046-50. doi: 10.1016/j.jaci.2004.08.036. PMID 15536408